CLINICAL TRIAL: NCT00324428
Title: The Effect of a 10-day Course of Transcranial Magnetic Stimulation on Abdominal Pain in Patients With Locally Advanced and Advanced Pancreatic Cancer, a Randomized Phase II Study.
Brief Title: TMS for the Treatment of Pancreatic Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005P000311; R03DK071851 (NIH)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Pain; Visceral Pain; Pancreatic Cancer
Keywords: TMS; Visceral Pain; Analgesia; Pancreatic Cancer; Cancer; Electric stimulation therapy; Electric stimulation; Pain; Safety
MeSH Terms: conditions — Pain; Visceral Pain; Pancreatic Neoplasms; Agnosia; Neoplasms | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial Magnetic Stimulation (TMS) (Experimental): This arm provides active 1Hz repetitive TMS (rTMS) applied to SII
  Interventions: Procedure: Transcranial Magnetic Stimulation
- Transcranial Magnetic Stimulation Sham (Sham Comparator): This arm provides sham 1Hz repetitive TMS (rTMS) applied to SII
  Interventions: Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — 1Hz repetitive transcranial magnetic stimulation for 10 days 26 minutes each day

SUMMARY:
This is a phase II study that aims to investigate prospectively a new therapy for a cohort of patients with chronic pain attributed to pancreatic cancer. The justification of this study is that the pain is the most important factor for the quality of life of these patients and rTMS has been shown to be significantly associated with pain improvement in patients with abdominal pain due to chronic pancreatitis. This therapeutic trial will be a 10-day, randomized, parallel-group design, double-blind, incomplete cross-over, placebo controlled clinical trial conducted at Beth Israel Deaconess Medical Center. The principal aim of this investigation is the study of pain after a therapeutic intervention. The primary outcome is pain reduction indexed by pain reduction and or analgesic intake reduction. The second aim of the study is to assess the safety this new treatment in patients with pancreatic cancer. The third aim of this study is to investigate whether rTMS treatment is associated with a change in the activity of right secondary somatosensory cortex using magnetic resonance spectroscopy. Because patients with locally advanced or advanced pancreatic cancer often require increasing doses of narcotic pain medications, such as morphine, oxycodone and fentanyl, in order to control their pain, adverse side effects are frequent observed in this population of patients. Therefore rTMS treatment might represent a new therapeutic approach that might be useful not only for pancreatic cancer but also to other types of cancer.

DETAILED DESCRIPTION:
The primary aim of this protocol is to investigate a possible novel treatment for visceral pain in patients with locally advanced or advanced pancreatic cancer. Pain is a major contributor to the poor quality of life in patients with pancreatic cancer. Most patients with locally advanced or advanced pancreatic cancer have abdominal pain that requires treatment with increasing doses of narcotic pain medication. The refractory nature of pancreatic cancer pain to pharmacologic therapy led us to hypothesize that one mechanism leading to pain in these patients is dysfunction of brain cortical regulation of visceral sensation. This notion is supported by the finding that deep electrical stimulation of the brain can produce pain relief in patients with intractable pain due to progressive cancers of various types. In addition, patients with pancreatitis, a non-malignant pancreatic condition causing chronic pain, can continue to experience disabling pain even after total pancreatectomy. These finding suggests that pain symptoms in pancreatic cancer can be sustained by a pancreas-independent, neural-based mechanisms in the brain.

Visceral sensation is processed in the secondary somatosensory area (SII). Therefore, pancreatic cancer pain may be sustained by dysfunction of SII rather than by local effects of the cancer alone. We hypothesize further, that dysfunction of SII is one of hyper-excitability. According to this hypothesis, suppression of SII activity may help control the pain in patients with pancreatic cancer and may provide synergy with pharmacologic treatment.

Temporary inhibition of SII activity can be obtained by a novel, non-invasive procedure called transcranial magnetic stimulation (TMS). TMS can suppress brain excitability beyond the duration of the direct application of TMS if appropriate stimulation parameters are utilized. This hypothesis is supported by a sham controlled, double blind pilot trial of 5 subjects with idiopathic chronic pancreatitis: active rTMS applied to SII resulted in significant pain improvement in three of the subjects while sham did not provide any benefit in any of these patients. Furthermore, recent evidence suggests that stimulation of other brain areas, such as the dorsolateral pre-frontal cortex, can modulate acute, experimentally invoked pain (Graff-Guerrero et al 2005).

We will rigorously test the hypothesis that pain due to pancreatic cancer is sustained by dysfunction of SII characterized by hyperexcitability through two specific aims:

1. The first aim of this study is to examine whether 1Hz repetitive TMS (rTMS) applied to SII for ten days during two consecutive weeks in patients with abdominal pain due to pancreatic cancer has an analgesic effect.

   1. The primary outcome for this aim is the difference in pain score level on the Visual Analogue Scale at Day 11 and at Day 28 compared to the week before rTMS. The null hypothesis is that there is no difference in pain score between pre and post-treatment.
   2. The secondary outcome for this aim is to assess the difference in the use of narcotics for pain control on Day 11 and Day 28 compared to Day 1. The null hypothesis is that there is no difference in narcotic use (in IV morphine equivalency units) between pre and post-treatment.
2. The second aim of the study is to assess the safety of rTMS in patients with pancreatic cancer.
3. The third aim of this study is to investigate whether rTMS treatment is associated with a change in the activity of right SII using magnetic resonance spectroscopy. Therefore we will compare the levels of these substances between the two different time points (baseline and post-treatment) and between left and right SII. We expect a decrease in the excitatory neurotransmitters levels (Glutamine - Glx) in the stimulated area as a result of the inhibitory rTMS.

SAFETY In a pilot study of chronic pancreatitis patients, no subject experienced adverse effects from a single session of rTMS. Subjects in an ongoing study of a 10-day course or rTMS in chronic pancreatitis patients also have not experienced adverse events (10 patients thus far). Fifteen-day courses of rTMS have been used for the treatment of various neuropsychiatric diseases without any complications if safety guidelines are carefully followed. We will adhere to the current safety recommendations for rTMS endorsed by the International Society for Transcranial Stimulation and the International Federation for Clinical Neurophysiology. Therefore, we hypothesize that the proposed rTMS protocol will be safe for our patient population.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic pancreatic cancer
* Abdominal pain attributable to pancreatic cancer that requires daily narcotic use
* Stable narcotic dosage the week before study entry
* A computed tomography of the abdomen within four weeks of study entry
* CA19-9 within four weeks of study entry
* ECOG Performance status >=3

Exclusion Criteria:

* Known brain metastasis
* Patients with major depression with suicidal risk
* Prior neurosurgical procedures
* History of epilepsy
* Previous head injury
* History of Stroke
* Abnormal neurological examination other than as signs of the condition studied in the present protocol
* Contraindication to TMS:

Implanted pacemaker;Medication pump;Vagal stimulator;Deep brain stimulator;Metallic hardware in the head or scalp: shrapnel, surgical clips, or fragments from welding;Signs of increased intracranial pressure

* TENS unit and ventriculo-peritoneal shunt
* Pregnancy

Unable to undergo a brain MR

* claustrophobia refractory to anxiolytics
* ferromagnetic metal in the body such as a prosthetic heart valve, a pacemaker, or a brain aneurysm clip).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pain (visual analog scale, CGI,PGA); Medication use (medication diary) | 1 year

SECONDARY OUTCOMES:
Safety (cognitive assessment - neuropsychological battery) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: TMS for the treatment of Chronic Pancreatitis — http://clinicaltrials.gov/ct/show/NCT00130052?order=1